CLINICAL TRIAL: NCT00029328
Title: Soluble Tumor Necrosis Factor Receptor: Enbrel (Etanercept) for the Treatment of Acute Pulmonary Dysfunction (Idiopathic Pneumonia Syndrome) Following Allogeneic Stem Cell Transplantation
Brief Title: Etanercept for Non-Infectious Lung Injury Following Bone Marrow Transplantation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: FD-R-2020-01; UMCC-0078;; FD-R-002020-01
Record Dates: First submitted 2002-01-10; First posted 2002-01-11 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2001-11

CONDITIONS: Respiratory Distress Syndrome, Adult; Bronchiolitis Obliterans; Pneumonia
Keywords: TNFR-Fc fusion protein; Stem Cell Transplantation; Transplantation, Homologous; Respiratory Function Tests
MeSH Terms: conditions — Respiratory Distress Syndrome; Bronchiolitis Obliterans; Pneumonia | interventions — Etanercept

INTERVENTIONS:
Drug: etanercept

SUMMARY:
The purpose of this study is to determine the effects of etanercept, and define the toxicity, when administered to patients with acute non-infectious lung injury (idiopathic pneumonia syndrome, IPS) and with subacute pulmonary dysfunction after allogeneic stem cell transplantation.

DETAILED DESCRIPTION:
Over the last 2 decades, allogeneic bone marrow transplantation (BMT) has emerged as an important treatment option for a number of malignant and non-malignant disorders. Unfortunately, pulmonary dysfunction remains a frequent and severe complication of allogeneic BMT. One of the main chemicals felt to cause lung damage is Tumor Necrosis Factor (TNF). Etanercept is an experimental drug that attempts to block TNF lung damage. Patients will undergo blood tests, x-rays, and a bronchoscopy with broncho-alveolar lavage prior to treatment with etanercept to check for infection. If no infection is evident after 24 hours, the etanercept will be started and administered twice weekly for 4 weeks by subcutaneous injection. There will be weekly blood tests and bronchoscopy after the last drug dose.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of acute idiopathic pneumonia syndrome (IPS) or sub-acute lung injury
* At least 1 year of age for IPS stratum
* At least 6 years of age for sub-acute lung injury stratum and able to perform formal pulmonary function testing
* At least 14 days since prior treatment with an investigational drug for graft-versus-host disease
* Previously treated with allogeneic stem cell or bone marrow transplantation for primary disease

Exclusion criteria:

* Documented evidence of active systemic or pulmonary infection
* Cardiogenic failure as cause of pulmonary dysfunction
* Known hypersensitivity to etanercept
* Currently receiving dialysis
* Currently receiving inotropic medications except dopamine
* Pregnant or nursing

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15
Dates: Start 2001-09; Study Completion 2003-09

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Cooke, M.D., Principal Investigator — University of Michigan, Ann Arbor, MI
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States